CLINICAL TRIAL: NCT05973591
Title: The Impact of Ivabradine on Left Ventricular Reverse Remodeling in Nonischemic Dilated Cardiomyopathy (NIDCM) on Current Medical Therapy Era
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-1665
Record Dates: First submitted 2023-07-16; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Dilated Cardiomyopathy; Ventricular Remodeling; Heart Failure, Reduced Ejection Fraction
MeSH Terms: conditions — Cardiomyopathy, Dilated; Ventricular Remodeling; Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- achieved HR ≥ 70 bpm without ivabradine: **Achieved HR : heart rate (HR) at 12 month follow up after the initiation of GDMT**
- achieved HR < 70 bpm without ivabradine: **Achieved HR : heart rate (HR) at 12 month follow up after the initiation of GDMT**
- achieved HR ≥ 70 bpm with ivabradine: **Achieved HR : heart rate (HR) at 12 month follow up after the initiation of GDMT**
- achieved HR < 70 bpm with ivabradine: **Achieved HR : heart rate (HR) at 12 month follow up after the initiation of GDMT**

SUMMARY:
In non-ischemic dilated cardiomyopathy (NIDCM), left ventricular reverse remodeling (LVRR) can be achieved through guideline-directed medical therapy (GDMT). LVRR is defined as an increase in left ventricular ejection fraction (LVEF) of more than 10% in heart failure patients with a baseline LVEF of 40% or less, or an increase in LVEF of more than 40% at follow-up, which is classified as heart failure with improved EF (HFimpEF) according to current guidelines. Several studies have examined the prevalence and predictors of LVRR in NIDCM. However, there is a lack of research on LVRR in the context of contemporary pharmacotherapy. Studies have demonstrated the beneficial effects of ivabradine in heart failure with reduced ejection fraction (HFrEF), improving patients' prognosis. A sub-study of the SHIFT trial indicated that ivabradine may also contribute to cardiac remodeling reversal in patients with HFrEF. However, there is limited evidence exploring the relationship between ivabradine and LVRR, particularly in the context of NIDCM.

Consequently, this study is a retrospective, multi-center cohort study aiming to evaluate the impact of ivabradine on LVRR in patients with NIDCM in the current era of medical therapy. Furthermore, by conducting this study, we aim to gain insights into the potential role of ivabradine in promoting LVRR in NIDCM patients receiving contemporary drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with non-ischemic dilated cardiomyopathy (NIDCM) by performing coronary artery imaging (coronary angiography, CT angiography, or SPECT scan) at the time of diagnosis of HFrEF
2. Sinus rhythm
3. Baseline LVEF of 40% or less (LVEF≤40%)
4. Patients containing baseline heart rate (HR)

   * In the Ivabradine group, baseline HR must be >75 bpm at the time of ivabradine dosing.

Exclusion Criteria:

1. Patients with confirmed ischemic cardiomyopathy (when stenosis of 75% or more of major coronary arteries is confirmed on coronary artery imaging or ischemic cardiomyopathy findings such as transmural LGE on cardiac MRI)
2. Heart failure with other etiologies (e.g., valvular heart disease, endocrine disease).
3. Previous recovery history of left ventricular systolic function (LVEF)
4. Cardiac resynchronization therapy (CRT) implantation
5. Persistent/permanent atrial fibrillation

7) Contraindication to the administration of ivabradine according to the Summary of Product Characteristics (SmPC)

* Hypersensitivity reactions
* Symptomatic bradycardia or resting heart rate < 75 bpm prior to treatment
* Cardiogenic shock, acute myocardial infarction, severe hypotension (< 90/50 mmHg), severe hepatic failure, sinus syndrome, atrial block, unstable or acute heart failure, pacemaker dependence (with pacing dominance), unstable angina, third degree atrioventricular block
* Cytochrome P450 3A4 inhibitors: Azole class antifungals (ketoconazole,itraconazole), Macrolide class antibiotics (clarithromycin, erythromycin per os, josamycin, telithromycin), HIV protease inhibitors (nelfinavir, ritonavir), nefazodone or any concomitant use with verapamil or diltiazem (moderate CYP3A4 inhibitors with heart rate reducing properties).

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with NIDCM with sinus rhythm
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of of LVRR in patients with NIDCM | at 12 months after the initiation of GDMT
  LVRR is characterized by an increase in left ventricular ejection fraction (LVEF) of more than 10% in heart failure patients with a baseline LVEF of 40% or less, or an increase in LVEF of more than 40% during follow-up, which is classified as heart failure with improved EF (HFimpEF). Furthermore, the initiation of guideline-directed medical therapy (GDMT) is defined as the timeframe for commencing treatment with an angiotensin-converting enzyme inhibitor (ACEi), angiotensin II receptor antagonist (ARB), or beta-blocker after the diagnosis of heart failure with reduced ejection fraction (HFrEF).

SECONDARY OUTCOMES:
Prevalence of LVRR in NIDCM at 8 months after initiation of GDMT | at 8 months after GDMT initiation
Extent of LVRR (measured by LVEDD/LVESD, LAVI, E/e' in echocardiography) in NIDCM at 8 and 12 months after GDMT initiation | at 8 and 12 months after GDMT initiation
Clinical course of LVRR in NIDCM | at 8 and 12 months after GDMT initiation
Effect of targeted HR (HF <60 or 70/min) on LVRR in NIDCM at 8 and 12 months after GDMT initiation | at 8 and 12 months after GDMT initiation
Effect of degree of change in HR before and after GDMT on LVRR in NIDCM at 8 and 12 months after GDMT initiation | at 8 and 12 months after GDMT initiation
Impact of GDMT on LVRR in NIDCM at 8 and 12 months after GDMT initiation | at 8 and 12 months after GDMT initiation
Prevalence of symptomatic bradycardia, syncope, or any other adverse events with Ivabradine | at 8 and 12 months after GDMT initiation

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Min Kang, Principal Investigator — Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No